CLINICAL TRIAL: NCT06584981
Title: Effect of PECS II, Parasternal and Serratus Plane Blocks on Postoperative Pain in MIDCAB Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Hasan Hüseyin KILIÇ, Hasan Huseyin Kilic, Hisar Intercontinental Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: HisarH
Record Dates: First submitted 2024-08-20; First posted 2024-09-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative; Coronary Artery Disease
MeSH Terms: conditions — Pain, Postoperative; Coronary Artery Disease | interventions — Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients who underwent block (Active Comparator): Patients who underwent pectoral nerve block (PECS II), parasternal and serratus plane blocks will be included in this group.
  Interventions: Procedure: pectoral nerve block (PECS II), parasternal and serratus plane blocks
- Patients who did not receive block (Other): Patients who were not given a block and received standard intravenous analgesics will be included in this group.
  Interventions: Other: analgesic

INTERVENTIONS:
Procedure: pectoral nerve block (PECS II), parasternal and serratus plane blocks — These block applications are performed under sterile conditions under the guidance of ultrasonography
  Arms: Patients who underwent block
Other: analgesic — Analgesia needs of patients who do not receive blockade are met with intravenous drugs.
  Arms: Patients who did not receive block

SUMMARY:
AIM: It was aimed to evaluate the effectiveness of pectoral nerve block (PECS II), parasternal and serratus plane blocks in postoperative analgesia in minimally invasive cardiac surgery (MIDCAB).

INTRODUCTION: The frequency of minimally invasive cardiac surgery has increased in recent years. With this method, Coronary artery bypass graft (CABG) operations can be performed without sternotomy. It is a beneficial method for early postoperative mobilization, early recovery and better aesthetic appearance. Since there is a surgical intervention between the ribs, pain control is important in these patients.

METHOD: In the preoperative evaluation of patients planned for CABG, PECS II, parasternal and serratus plane blocks are routinely recommended for postoperative pain control. Consent for the procedure is obtained from patients who accept this procedure. After induction and before the surgical incision, these block applications are performed under sterile conditions under the guidance of ultrasonography. Standard intravenous analgesic agents are applied to our patients who do not accept block applications. The hospital core system files of our patients who underwent cardiac surgery with minimally invasive intervention in our hospital between January 1, 2021 and December 31, 2021 will be scanned retrospectively. Patients with and without block application will be divided into two groups. From our patients' files; Demographic data, extubation time, drain site and incision site pain at the 1st, 2nd, 4th, 12th, 24th, 48th and 72nd hours after extubation will be noted. In addition, it will be noted whether there is a need for additional rescue analgesia in cases where block is performed. The data obtained will be evaluated statistically and the results will be published in national or international scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 and over
* Patients who underwent MIDCAB surgery

Exclusion Criteria:

* Patients under 18 years of age
* Patients who did not undergo MIDCAB surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Analgesic efficiency | drain site and incision site pain at the 1st, 2nd, 4th, 12th, 24th, 48th and 72nd hours after extubation will be noted

CONTACTS AND LOCATIONS:
Locations (1):
- Hisar Intercontinental Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Gautam S, Pande S, Agarwal A, Agarwal SK, Rastogi A, Shamshery C, Singh A. Evaluation of Serratus Anterior Plane Block for Pain Relief in Patients Undergoing MIDCAB Surgery. Innovations (Phila). 2020 Mar/Apr;15(2):148-154. doi: 10.1177/1556984520908962. PMID 32352903
- [Result] Morimoto Y, Sakata M, Ohno A, Maegawa T, Tajima S. [Effects of bofu-tsusho-san, a traditional Chinese medicine, on body fat accumulation in fructose-loaded rats]. Nihon Yakurigaku Zasshi. 2001 Jan;117(1):77-86. doi: 10.1254/fpj.117.77. Japanese. PMID 11233300
- [Result] Moll V, Ward CT, Jabaley CS, O'Reilly-Shah VN, Boorman DW, McKenzie-Brown AM, Halkos ME, Prabhakar A, Pyronneau LR, Schmidt PC. Erector Spinae Regional Anesthesia for Robotic Coronary Artery Bypass Surgery Is Not Associated With Reduced Postoperative Opioid Use: A Retrospective Observational Study. J Cardiothorac Vasc Anesth. 2021 Jul;35(7):2034-2042. doi: 10.1053/j.jvca.2020.09.112. Epub 2020 Sep 20. PMID 33127286